CLINICAL TRIAL: NCT07124754
Title: Development and Validation of a Multimodal Artificial Intelligence Model for Predicting Lymph Node Metastasis in T1 Gastric Cancer and Its Impact on Physician Diagnostic Performance
Brief Title: Multimodal Deep Learning for Lymph Node Metastasis Prediction and Physician Performance Assessment in T1 Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: Qun Zhao (Other)
Responsible Party: Sponsor-Investigator, Qun Zhao, Professor, Hebei Medical University
Organization: Hebei Medical University (Other)
Other Study IDs: GC-RAD-AI-2025-04
Record Dates: First submitted 2025-08-03; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: T1 Gastric Cancer Lymph Node Metastasis Early Gastric Cancer Artificial Intelligence-Assisted Diagnosis Multimodal Data Integration
Keywords: T1 Gastric Cancer Lymph Node Metastasis Early Gastric Cancer Artificial Intelligence-Assisted Diagnosis Multimodal Data Integration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Multimodal Artificial Intelligence Diagnostic Model for Lymph Node Metastasis in T1 Gastric Cancer — This intervention involves the use of a custom-built artificial intelligence (AI) diagnostic model that integrates multimodal data-including clinical variables, histopathological features, and imaging data-to predict lymph node metastasis in patients with T1-stage gastric cancer.
  The model provides risk probability scores and classification outputs that assist physicians in diagnostic decision-making.
  The AI system will be compared with physician performance at different levels of experience (resident, attending, senior) to assess its impact on diagnostic accuracy and clinical decision support.

SUMMARY:
This study aims to develop and validate an artificial intelligence (AI) model that integrates clinical, pathological, and imaging data to predict the presence of lymph node metastasis (LNM) in patients with T1-stage gastric cancer.

The study will also compare the diagnostic performance of physicians with and without AI assistance, including clinicians with varying levels of experience.

The goal is to improve early decision-making and support more personalized treatment strategies for patients with early gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

Age 18 years or older

Histologically confirmed primary gastric adenocarcinoma

Clinical stage T1 (T1a or T1b) confirmed by endoscopy and imaging

Undergoing radical gastrectomy with lymph node dissection

Preoperative data available: clinical variables, CT imaging, and pathology slides

Written informed consent provided

Exclusion Criteria:

History of other malignancies within the past 5 years

Received neoadjuvant chemotherapy or radiotherapy

Incomplete clinical or pathological data

Poor quality or missing CT or histopathology images

Patients with distant metastasis (M1) at diagnosis

Inability or refusal to provide informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with T1-stage gastric adenocarcinoma who undergo radical gastrectomy with lymph node dissection at participating centers. Participants must have available preoperative clinical, imaging, and pathological data for AI model input and postoperative histopathological confirmation of lymph node status.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of the AI Model for Predicting Lymph Node Metastasis in T1 Gastric Cancer | Immediately after surgery (within 7 days postoperatively, based on final pathological report)
Diagnostic Accuracy of the AI Model for Predicting Lymph Node Metastasis in T1 Gastric Cancer | At the time of final pathological diagnosis (typically within 3-7 days after surgery)

CONTACTS AND LOCATIONS:
Locations (1):
- the Fourth Hospital of Hebei Medical University, Shijiazhuang, None Selected, China

IPD SHARING:
Plan to Share IPD: Undecided